CLINICAL TRIAL: NCT03675711
Title: Midline Catheter and Its Impact on Central Lines Removal in ICU
Acronym: MIDREA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment problem
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD 037-18
Record Dates: First submitted 2018-09-04; First posted 2018-09-18 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Vascular Access Device

STUDY DESIGN:
Intervention Model Description: supportive care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midline Catheter (Active Comparator): Pt. will receive midline catheters.
  Interventions: Device: Midline
- Standard Peripheral venous Catheter (Active Comparator): Pt. will receive a standard Peripheral venous catheter
  Interventions: Device: PVC

INTERVENTIONS:
Device: Midline — Patient will receive a Midline catheter within 48h after disappearance of indication for CVC
  Arms: Midline Catheter
Device: PVC — Patient will receive a standard PVC within 48h after disappearance of indication for CVC
  Other Names: Conventional catheterization
  Arms: Standard Peripheral venous Catheter

SUMMARY:
The study will evaluate 2 strategies to remove central venous catheter (CVC): in one part, the insertion of a midline catheter and in the other part, the conventional insertion of peripheral venous catheter (PVC)

DETAILED DESCRIPTION:
Patients will be randomised when the last indication for CVC has disappeared, which means parenteral nutrition or vasopressors administration.

They will be randomised either in the midline group or in the PVC group.

* In the midline group, a midline catheter will try to be inserted before the 48th hour after last indication for CVC disappeared.
* In the PVC group: a PVC will try to be inserted before the 48th hour after last indication for CVC disappeared.

If successful, CVC will then be removed. If not, a PVC will try to be inserted daily till success or worthlessness of a venous line or death.

The presence of a CVC will be assessed at the 96th hour after disappearance of last CVC indication.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* admitted to ICU since at least 48h
* with a perfusion CVC inserted
* requiring or having required invasive mechanical ventilation
* lack of formal indication to CVC maintenance (weaning of vasopressors and/or parenteral nutrition) since at least 24 hours
* indication to maintain a venous access

Exclusion Criteria:

* Lack of patient or next of kin consent
* Personnel for insertion of midline catheter not available
* Admission in ICU before study start
* Admission following a transfer from another ICU
* Patient with an implantable port or a peripherally inserted central catheter (PICC Line)
* Known intolerance to components of study Midline device
* Past history of irradiation of insert area of midline catheter
* Past history of bilateral axillary lymph node dissection
* Pre-existing skin infection on upper limb
* Patient with a treatment-limitation decision
* Patient admitted after cardiac arrest with non-shockable rhythm
* Moribund
* Pregnancy, breastfeeding woman
* Patient under legal guardianship
* Patient hospitalized without consent and/or deprived of liberty by court's decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
% of patient with a successful Removal of CVC at the 96th hour after disappearance of last indication for CVC | H96 : 96th hour after disappearance of last indication for CVC
  A successful removal of CVC is defined as
  * success of midline/PVC insertion at H96 and consequently CVC removal
  * and no necessity for insertion of a new CVC within the 96 first hours

SECONDARY OUTCOMES:
Total number of puncture required for the insertion of a peripheral catheter | until 28 days after randomisation
Total number of peripheral catheter used | until 28 days after randomisation
Number of new CVC inserted | until 28 days after randomisation
Time consumption | until 28 days after randomisation
  Total time of catheterisation, (measured from the entrance in patient room, to the exit)
Number of blood culture for research of catheter-related bloodstream infection (CRBSI) | until 28 days after randomisation
CVC dwell time | from disappearance of CVC indication to last CVC removal or 28 days after randomisation if still in place
  Time of central catheter duration (hours)
Number of CVC colonized for per 1000 CVC /days | until 28 days after randomisation
Number of CVC-associated bacteremia | until 28 days after randomisation
Number of peripheral catheter-associated bacteremia | until 28 days after randomisation
ICU length of stay | Until discharge from ICU, an expected average of 12 days
Hospital length of stay | Until discharge from hospital, an expected average of 20 days
  Hospital stay in medical and surgical unit (no follow-up and rehabilitation care unit or long stay)
ICU mortality | Until discharge from ICU, an expected average of 12 days
hospital mortality | Until discharge from hospital, an expected average of 20 days
  mortality in medical and surgical unit (no SSR or long stay)

OTHER OUTCOMES:
Colonization of Midline at removal | until removal,an expected average of 10 days after insertion
  swabbing will be performed at catheter removal and its tips will be also analyzed
Colonization of skin at insert point of Midline catheter | until 28 days after randomisation
  swabbing will be performed at every change of dressing
Thrombosis at Midline removal | until removal in ICU,an expected average of 10 days after insertion
  thrombosis will be checked by ultrasound-echography if midline is removed in ICU

CONTACTS AND LOCATIONS:
Overall Officials: angelina robert, Principal Investigator — CHD vendee
Locations (1):
- Centre Hospitalier Departemental Vendée, La Roche-sur-Yon, France